CLINICAL TRIAL: NCT04315220
Title: Effectiveness of Core Stability Training in Improving Postural Stability and Foot Pressure Distribution in Overweight Children: A Randomized Controlled Trial
Brief Title: Corestability Training in Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Collaborators: Maharishi Markandeshwar International School (Unknown)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/2020; U1111-1249-8305 (Other: Universal Trial Number (UTN) by WHO ICTRP)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Childhood Obesity; Child Obesity; Children, Only
Keywords: Noncommunicable disease; Balance; Posture; Childhood obesity; Overweight
MeSH Terms: conditions — Pediatric Obesity; Noncommunicable Diseases; Overweight

STUDY DESIGN:
Intervention Model Description: Two group pre-test post-test design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Core stability training (CST)) (Experimental): Core stability training (CST) consists of two levels: level 1- Mat exercises (includes abdominal muscle contraction, bridging,cat stretch,single leg circle and superman) and level 2- Swiss ball exercises (includes abdominal muscle contraction, bridging and squatting by using therapy ball).
  There will be three sets of 15 repetitions of each exercises. The first set will consist of 10 seconds hold period, follow by 12 seconds hold in second set and 15 seconds hold in third set respectively. The entire session will last for approximately 30 minutes.
  Interventions: Other: Corestability training
- Control group (Active Comparator): Will not receive any kind of training.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: Corestability training — Level -1: Mat exercises
  Abdominal muscle contraction,bridging,cat stretch,single limb circle and superman.:
  Level- 2: Swiss Ball Exercises Abdominal contraction,bridging and squats.
  Arms: Experimental group (Core stability training (CST))
Other: No Intervention — No Intervention
  Arms: Control group

SUMMARY:
A total of 52 overweight children aged between eight and sixteen years will be recruited by criterion based purposive sampling to participate in the two groups pretest post test randomized clinical study. Random allocation of the eligible subjects for treatment will be done by the block randomization method with matrix of thirteen rows and four columns (13x4). The subject will be allotted to the group randomly, based on the chit selected by the person other the primary researcher.Once the block is filled, the next row block will be opened. Thus equal distribution of overweight children in the each group will be ensured.

Group A will be receiving actual core stability training (Level 1 - Mat exercises and Level 2 - Swiss Ball exercises) for 6 weeks with a frequency of three sessions per week.Group B will receive no training. Each session will last for 30 minutes of duration. The static and dynamic balance, foot pressure distribution and core strength will be assessed at the baseline and at the end of the treatment sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Children of age 8- 16 years old.
2. Both Boys and Girls.
3. Child with BMI-for-age percentile growth between 85th to less than 95th percentile.

Exclusion Criteria:

1. Uncooperative participants.
2. Upper or lower limb fracture or injury in recent 6 months.
3. Any musculoskeletal or neurological disorder affecting core strength and balance.
4. Refuse to participate because not able to understand the researcher instructions.
5. Unable to attend the whole sessions during the research period.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Foot pressure distribution | change from baseline and six weeks
  All overweight children will be asked to walk barefoot along a 5-.metre walkway using Harris mat pressure distribution platform which will be placed on a firm, level surface, in the centre of walkway. Children will be ensured to step on the Harris mat without pause, first with one foot and then repeat the same procedure with the other foot at constant speed. Foot markings then analyzed by using
Single limb stance | change from baseline and six weeks
  The children will be instructed to stand on the dominant leg with non dominant leg flexed to 90 degree, and maintain the position. The test will be performed first with eyes open and then with the eyes closed. The time for which participant will be able to maintain balance will be recorded
Y- reach set | change from baseline and six weeks
  The participant will stand on one foot in the center of the Y with the most distal aspect of the toes just behind the starting line. While maintaining single-leg stance, the balance will be tested in the anterior, postero-medial and postero-lateral direction with reach foot. The reach distance in all the three directions will be noted.
Core Strength | change from baseline and six weeks
  The core strength will be measured with the Chattanooga Pressure Biofeedback Unit. The device will be placed under the lumbar spine in crook lying and inflated to a baseline of 40 mmHg. The participants will be instructed to perform drawing-in maneuver on the verbal instructions, maintain it for 10 sec. The change in pressure will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Kanu Goyal, BPT, DOMTP, Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Asir J Samuel, MPT, PhD, Study Chair — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (1):
- Kanu Goyal, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Detail protocol will be published highlighting methods, statistical plan and Informed consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once (Before the start start)
Access Criteria: Mendeley data Upload